CLINICAL TRIAL: NCT04281030
Title: Improving Health Outcomes of Migraine Patients Who Present to the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-00548 - 2; 1K23AT009706-01 (NIH)
Record Dates: First submitted 2019-12-26; First posted 2020-02-21 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (PMR) Therapy (Experimental): After the PMR APP is loaded onto the subject's smartphone, the subject will perform PMR in the ED and discuss the optimal time and place to practice PMR at home. All subjects will be asked to keep records of headache occurrence, side effects, compliance, and medication changes on the APP.
  Interventions: Behavioral: PMR (Progressive muscle relaxation therapy)
- Monitored Usual Care (MUC) (Active Comparator): Subjects will be given general educational information consisting of basic migraine information such as evidence-based ways to treat migraine: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently. Any migraine treatment decisions on discharge will be left up to the ED attending. The research coordinator (RC) will load the APP onto the subjects' smart phones but the PMR component will be blocked on the version of the APP that the MUC subjects receive. All subjects will be asked to keep records of headache occurrence, side effects, compliance, and medication changes on the APP.
  Interventions: Behavioral: Monitored Usual Care (MUC)

INTERVENTIONS:
Behavioral: PMR (Progressive muscle relaxation therapy) — Technique for learning to monitor and control the state of muscular tension. The relaxation therapy should take about 20 minutes a day.
  Arms: Progressive Muscle Relaxation (PMR) Therapy
Behavioral: Monitored Usual Care (MUC) — Subjects will be given basic migraine information such as evidence-based ways to treat migraine: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently.
  Arms: Monitored Usual Care (MUC)

SUMMARY:
This is a pilot feasibility acceptability study to examine the impact of smartphone-based progressive muscle relaxation (PMR) on migraine quality of life, frequency, intensity, and disability. Feasibility is measured by: a) Proportion of patients who enrolled in the study/were recruited for the study, b) Number of days PMR practiced/week as determined with the backend analytics in the RELAXaHEAD app, c) Minutes/day spent doing PMR, d) Reasons for non-adherence. Acceptability is measured by: a) Satisfaction using Likert scale questions on RELAXaHEAD usability, content, and functionality b) Willingness to repeat a similar treatment intervention in the future (Definitely No/Probably No/Unsure/Probably Yes/ Definitely Yes) c) Attrition. In addition, whether use of electronically based PMR introduced in the emergency department (ED) improves migraine quality of life (MSQv2) and migraine related disability (MIDAS) at 3 months post ED-discharge (or post enrollment date if recruited post ED discharge) compared to those who are not introduced to PMR will be assessed. All participants will be asked to track their headache frequency and intensity using our smartphone application (app) and will be asked to complete migraine quality of life assessments and migraine related disability at follow-up.

DETAILED DESCRIPTION:
While explaining the study, potential participants will be assured that they will receive all of the medication for their acute headache that they would otherwise receive. Once consented, participants will be randomized to PMR therapy or monitored usual care (MUC). Participants will be told that either group is being tested as an enhancement to the care they typically get in the ED for headache. (At the end, they will be informed which group they were in.) The study team will collect participants' health histories (biologic variables) and baseline data in REDCap, download the app onto subjects' smartphones, and conduct the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Meets migraine criteria and has 4+ headache days a month

Exclusion Criteria:

* Patients who have had Cognitive Behavioral Therapy, Biofeedback or other Relaxation Therapy in the past year
* Cognitive deficit or other physical problem with the potential to interfere with behavioral therapy
* Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record
* Unable or unwilling to follow a treatment program that relies on written and audio recorded materials
* Not having a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Will be provided upon request

REFERENCES:
- [Derived] Minen MT, Seng EK, Friedman BW, George AD, Fanning KM, Bostic RC, Powers SW, Lipton RB. Smartphone-Based Muscle Relaxation for Migraine in the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2534221. doi: 10.1001/jamanetworkopen.2025.34221. PMID 41100087

RESULTS

PARTICIPANT FLOW:
Groups:
- Progressive Muscle Relaxation (PMR) Therapy: After the Progressive Muscle Relaxation (PMR) APP is loaded onto the subject's smartphone, the subject will perform PMR in the emergency department (ED) and discuss the optimal time and place to practice PMR at home. All subjects will be asked to keep records of headache occurrence, side effects, compliance, and medication changes on the APP.
  PMR (Progressive muscle relaxation therapy): Technique for learning to monitor and control the state of muscular tension. The relaxation therapy should take about 20 minutes a day.
Period: Overall Study
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Started | 56 | 56
Participants Allocated to Intervention | 54 | 54
Completed | 46 | 48
Not Completed | 10 | 8
Not completed — Technology issues prevented participant from receiving intervention | 2 | 2
Not completed — Participant excluded from analysis as they did not meet criteria of MIDAS score > 5 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Monitored Usual Care (MUC): Subjects will be given general educational information consisting of basic migraine information such as evidence-based ways to treat migraine: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently. Any migraine treatment decisions on discharge will be left up to the ED attending. The RC will load the APP onto the subjects' smart phones but the PMR component will be blocked on the version of the APP that the MUC subjects receive. All subjects will be asked to keep records of headache occurrence, side effects, compliance, and medication changes on the APP.
  Monitored Usual Care (MUC): Subjects will be given basic migraine information such as evidence-based ways to treat migraine: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently.
- Total: Total of all reporting groups
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC) | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [25 to 43] | 36 [28 to 46] | 33.5 [26 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 9 | 8 | 17
  Other Gender | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 10 | 26
  Not Hispanic or Latino | 29 | 37 | 66
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 23 | 27 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Migraine Disability Assessment Scale (MIDAS) Score
Description: 5-item self-administered questionnaire designed to quantify headache-related disability over a 3-month period. For each item, participants indicate the number of days over the past three months that migraine limited their ability to participant in specific activities.
  The score is the sum responses. Scores are classified as follows:
  * 0 to 5 = Little or no disability (MIDAS Grade I)
  * 6 to 10 = Mild disability (MIDAS Grade II)
  * 11 to 20 = Moderate disability (MIDAS Grade III)
  * 21-40 = Severe disability (MIDAS Grade IV-A)
  * Greater than 40 = Very severe disability (MIDAS Grade IV-B)
Time Frame: Baseline, Month 3 Post-Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Number analyzed (Participants) | 34 | 35
score on a scale | -25.1 (29.6) | 6.9 (59.6)

2. Secondary Outcome: Number of Headache Days Based on MIDAS
Description: Information from the Migraine Disability Assessment Scale (MIDAS) questionnaire will be used to calculate the number of headache days at baseline.
Time Frame: Baseline
Measure: Mean (Inter-Quartile Range); unit: Headache Days
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Number analyzed (Participants) | 46 | 48
Headache Days | 14 [6 to 20] | 10 [5 to 16]

3. Secondary Outcome: Change in Migraine-Specific Quality of Life Questionnaire-Version 2 (MSQv2) - Role Function Restrictive (RFR) Domain Scores
Description: The MSQv2 is a 14-item self-assessment of how migraines affect a patient's life. 7 of the items assess the Role Function-Restrictive (RFR) Domain, which measures the functional impact of migraine through limitations on daily social and work activities.
  Items are ranked on 6-point Likert scale, where: 1 = None of the time; 2 = A little bit of the time; 3 = Some of the time; 4 = A good bit of time; 5 = Most of the time; and 6 = All of the time.
  The raw dimension score is computed as a sum of item responses and rescaled on a 0-100 scale; higher scores indicate better quality of life.
Time Frame: Baseline, Month 3 Post-Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Number analyzed (Participants) | 34 | 35
score on a scale | 18.1 (18.1) | 18.7 (26.8)

4. Secondary Outcome: Change in MSQv2 - Emotional Function (EF) Domain Scores
Description: The MSQv2 is a 14-item self-assessment of how migraines affect a patient's life. 3 of the items assess the Emotional Function (EF) Domain, which measures the emotional impact of migraine.
  Items are ranked on 6-point Likert scale, where: 1 = None of the time; 2 = A little bit of the time; 3 = Some of the time; 4 = A good bit of time; 5 = Most of the time; and 6 = All of the time.
  The raw dimension score is computed as a sum of item responses and rescaled on a 0-100 scale; higher scores indicate better quality of life.
Time Frame: Baseline, Month 3 Post-Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Number analyzed (Participants) | 34 | 35
score on a scale | 26.5 (26.5) | 19.8 (38.5)

5. Secondary Outcome: Change in MSQv2 - Role Function Preventive (RFP) Domain Scores
Description: The MSQv2 is a 14-item self-assessment of how migraines affect a patient's life. 4 of the items assess the Role Function-Preventive (RFP) Domain, which measures the impact of migraine through prevention of daily work and social activities
  Items are ranked on 6-point Likert scale, where: 1 = None of the time; 2 = A little bit of the time; 3 = Some of the time; 4 = A good bit of time; 5 = Most of the time; and 6 = All of the time.
  The raw dimension score is computed as a sum of item responses and rescaled on a 0-100 scale; higher scores indicate better quality of life.
Time Frame: Baseline, Month 3 Post-Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
Number analyzed (Participants) | 34 | 35
score on a scale | 16.9 (16.9) | 11.3 (25.9)

ADVERSE EVENTS:
Description: Adverse events, serious adverse events, and all-cause mortality were not assessed among participants in this study, as minimal to no risk was expected for participants in the study.
Groups:
- Monitored Usual Care (MUC): Subjects will be given general educational information consisting of basic migraine information such as evidence-based ways to treat migraines: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently. Any migraine treatment decisions on discharge will be left up to the ED attending. The RC will load the APP onto the subjects' smart phones but the PMR component will be blocked on the version of the APP that the MUC subjects receive. All subjects will be asked to keep records of headache occurrence, side effects, compliance, and medication changes on the APP.
  Monitored Usual Care (MUC): Subjects will be given basic migraine information such as evidence-based ways to treat migraine: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently.
Arm/Group | Progressive Muscle Relaxation (PMR) Therapy | Monitored Usual Care (MUC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT04281030/Prot_SAP_000.pdf